CLINICAL TRIAL: NCT00266994
Title: HTRS TE Registry (ThromboEmbolism Registry): Prospective Registry of Demographic and Clinical Data for Patients With Thromboembolic Disease
Brief Title: HTRS TE Registry (ThromboEmbolism Registry)
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Hemophilia and Thrombosis Research Society (Unknown)
Responsible Party: Principal Investigator, Bryce A. Kerlin, PI, Nationwide Children's Hospital
Other Study IDs: 05-00343; 502305
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Thromboembolism
Keywords: Thrombosis
MeSH Terms: conditions — Thromboembolism; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The TE Registry is a multi-institutional bioinformatics database for the collection of data relevant to TE. Participating HTRS affiliated study centers may enroll patients and enter data in the TE Registry by completing enrollment and data entry forms and transmitting them to the study center. The purpose of this study is to improve our understanding of the epidemiology, pathophysiology, and outcome of patients suffering from thromboembolism (TE) events.

The initial objectives of the registry are:

* Evaluate the epidemiology and clinical characteristics of known prothrombotic risk factors in persons with TE.
* Identify the frequency and nature of complications associated with TE and its treatment.
* Describe the phenotypes and complications seen in persons with multiple molecular risk factors for TE.
* Compare the epidemiology, clinical characteristics, and complications seen in patients with and without known risk factors for TE.

DETAILED DESCRIPTION:
Hereditary defects that predispose to thromboembolism (TE) and its complications afflict 5-8% of the U.S population. Annually, ~60,000 Americans die from TE and half of the survivors suffer long-term morbidity. Despite these staggering statistics, little is known about the clinical characteristics or epidemiology of the inherited risk factors for TE. Less is known regarding the acquired risk factors or the phenotype of TE in persons with multiple risk factors, yet preliminary data suggest that as many as 10% of patients may have multiple risk factors.

Data from several studies, primarily involving adult subjects, shows that in a population of consecutively studied thrombosis patients, that one of the five most common inherited predispositions will occur in ~33.8%. Antithrombin (AT) is the least common (~1.9%) of these, while Factor V Leiden (FVL) is the most common (~18.8%). Most children who suffer from TE have indwelling catheters to assist therapy of underlying medical conditions, or are sick neonates. Thus, the contribution of molecular risk factors in children is largely unknown, with the exception of sparse retrospective data.

The TE Registry may help clearly define the clinical phenotype, epidemiology, and complications seen in patients with TE associated with known molecular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be enrolled at the time of their FIRST thromboembolic event. Ideally, patients should be enrolled within three months of the diagnosis of an eligible event.
* Deep Venous, Arterial, or Intra-Cardiac Thrombosis
* Pulmonary Thromboembolism AND:

  * Must have evidence of Venous Thrombosis on imaging studies -OR-
  * Must have elevated Quantitative or Semi-Quantitative D-dimer level (as defined by local laboratory technology/normal ranges)
* Arterial Thromboembolism (with imaging evidence of thrombus source)
* Stroke (Cerebral Vascular Accident) AND age < 20 years. Stroke is defined as a completed stroke with symptoms persisting for > 24 hours and radiographic evidence of infarction by Computed Tomography or Magnetic Resonance Imaging. Transient Ischemic Attacks (TIA) are NOT eligible for this registry.
* Myocardial Infarction AND age <20 years. Must have elevated cardiac enzymes (CK and/or Troponin) and Electrocardiographic (EKG) evidence meeting the local standard for diagnosis. Angina is NOT eligible for this registry.

Exclusion Criteria:

* Bleeding disorders
* Transient Ischemic Attack(s) (TIA)
* Sickle Cell Disease
* Mitochondrial Encephalopathy, Lactic Acidosis, and Stroke-Like Episodes (MELAS)
* Ornithine Transcarbamylase Deficiency
* Homocystinuria
* Other metabolic disorders known to be associated with Stroke
* Hemorrhagic Stroke
* Bacterial Endocarditis
* Microangiopathic Hemolytic Anemias (Thrombotic Thrombocytopenic Purpura or Hemolytic Uremic Syndrome)
* Patients greater than or equal to 20 years of age with Stroke or Myocardial Infarction (in order to limit confounding cardiovascular risk factors)
* Angina

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients diagnosed with a thromboembolic event at any of the participating study centers will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2760 (Actual)
Dates: Start 2005-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Observation | 2 years
  Observational cohort study - no primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bryce A Kerlin, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States